CLINICAL TRIAL: NCT06340477
Title: Effect of Thoracic SNAGS on Vitals Among Individuals With Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mahnoor Arif/ REC -01802
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Neck Pain
Keywords: Forward head posture; vitals; SNAGs; craniovertebral angle
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic SNAGs with conventional therapy (Experimental): Thoracic (T1- T5) SNAGs 3 repetitions x 1 set, 2 days/week Hot pack for 10 minutes Stretching of upper trapezius, levator scapulae, 5 reps x 1 set x 15 sec hold 2 days/week and Pectoralis Major 10 reps x 1 set x 10 sec hold
  Strengthening of deep neck flexors and shoulder retractors (rhomboids) 10 reps x 1 set x 10 sec hold 2 days/week 2 days/week
  Interventions: Other: Thoracic SNAGs with conventional therapy
- Conventional therapy (Other): Hot pack for 10 minutes Stretching of upper trapezius, levator scapulae, 5 reps x 1 set x 15 sec hold 2 days/week and Pectoralis Major 10 reps x 1 set x 10 sec hold
  Strengthening of deep neck flexors and shoulder retractors (rhomboids) 10 reps x 1 set x 10 sec hold 2 days/week 2 days/week
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: Thoracic SNAGs with conventional therapy — Thoracic (T1- T5) SNAGs 3 repetitions x 1 set, 2 days/week Hot pack for 10 minutes Stretching of upper trapezius, levator scapulae, 5 reps x 1 set x 15 sec hold 2 days/week and Pectoralis Major 10 reps x 1 set x 10 sec hold
  Strengthening of deep neck flexors and shoulder retractors (rhomboids) 10 reps x 1 set x 10 sec hold 2 days/week 2 days/week
  Arms: Thoracic SNAGs with conventional therapy
Other: conventional therapy — Hot pack for 10 minutes Stretching of upper trapezius, levator scapulae, 5 reps x 1 set x 15 sec hold 2 days/week and Pectoralis Major 10 reps x 1 set x 10 sec hold
  Strengthening of deep neck flexors and shoulder retractors (rhomboids) 10 reps x 1 set x 10 sec hold 2 days/week 2 days/week
  Arms: Conventional therapy

SUMMARY:
To determine how vitals (heart rate, blood pressure, respiratory rate, oxygen saturation) and craniovertebral angle will be affected by thoracic SNAGs in individuals with forward head posture.

DETAILED DESCRIPTION:
Forward head posture (FHP) leads to abnormal activation of neck muscles. This leads to respiratory complications and changes in blood pressure. Due to regional interdependence Upper thoracic spine can restrict the movement of cervical spine Thoracic spine is is closely related to Sympathetic nervous system. T1-T5 spinal sympathetic neurons provide sympathetic innervation to the vessels that supply to the heart tissues and upper portion of the body. Thus, thoracic mobilization can regulate main body vitals as well as other visceral activities that maintain homeostasis

There is a manual therapy technique called sustained natural apophyseal glides (SNAGs) in which patient performs active movements along with the passive movements performed by the physiotherapist. It not only has biomechanical efficacy which includes pain reduction and improvement in ROM, but it also has neurophysiologic effects. Previous studies lack to provide how thoracic SNAGs can affect vitals. Thus, this study aims to determine the effect of thoracic SNAGs on vital signs, including heart rate, blood pressure, respiratory rate, and oxygen saturation . Furthermore, this research will add to growing body of knowledge that how thoracic SNAGs can influence the correction of forward head posture

ELIGIBILITY:
Inclusion Criteria:

* Both males and females
* Age 30-50yrs.
* Craniovertebral angle <50°
* Mild to moderate neck pain ranging between 3-6 on NPRS scale.
* Individuals with normal vitals:
* Heart rate (60-100 beats per minute)
* Respiratory rate (12-20 breaths per minute)
* Systolic BP (100- 139mmHg)(30).
* Diastolic BP (70-89 mmHg) (30).
* Oxygen saturation ≥96%

Exclusion Criteria:

* History of cervical/thoracic spine surgery
* Cardiopulmonary disorder or Hypertension ≥140/90mmHg (30).
* Vertebral instability
* Smokers
* Any infection or tumor

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Aneroid sphygmomanometer | 4 weeks
  Aneroid sphygmomanometer has more sensitivity and specificity (86.7% and 98.7%) than a digital device (80% and 67.7%) in the measurement of blood pressure, so it is considered to be more precise than a digital one
Pulse oximeter | 4 weeks
  Hypoxemia can be ruled out by pulse oximeter. It has high reliability and validity for heart rate calculation with ICC> 0.93 in healthy individuals.
Respiratory rate | 4 weeks
  Respiratory rate or the number of breaths per minute is defined as one breath to each movement of air in and out of the lungs. In general, the respiratory rate for an adult sits between 12 and 20 breaths per min. 60second count is more accurate than short duration i.e 15 and 30 second

SECONDARY OUTCOMES:
NPRS (Numeric Pain Rating Scale) | 4 weeks
  Numeric Pain Rating Scale (NPRS) measures the subjective intensity of pain. The NPRS is an eleven-point scale from 0 to 10. "0" = no pain and "10" = the most intense pain imaginable while the NPRS exhibited moderate reliability (ICC = 0.27-0.84)
Inclinometer | 4 weeks
  An inclinometer is used to measure the range of motion (ROM) of joints. It has a housing that contains a sensor. The sensor is sensitive to gravity and measures the angle of the housing. The angle is then displayed on a digital display or a dial. It is placed on the joint and then move the joint through its range of motion. The angle of the inclinometer will change as the joint moves. The maximum angle reached is the ROM of the joint. ICC values of inclinometer range between 0.89-0.94 in measuring cervical range of motion including flexion, extension, lateral flexion, and rotation; making it a reliable tool.
Photogrammetric method for craniovertebral angle | 4 weeks
  FHP can be measured by craniovertebral angle which measures natural head neck posture in the sagittal plane and is determined by the intersection of a line extending from tragus of ear to C7 and horizontal line passing through C7. Kinovea software will be used for measurement of Cranio vertebral angle. Inter-rater reliability ranged from an intraclass correlation coefficient value of 0.95 to 0.98, whereas the intrarater reliability ranged from an intraclass correlation coefficient value of 0.98 to 0.99

CONTACTS AND LOCATIONS:
Overall Officials: maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No